CLINICAL TRIAL: NCT07014904
Title: "Cytotoxic T Lymphocyte-Associated Antigen-4 (CTLA-4) Gene Single-nucleotide Polymorphism in Primary Immune Thrombocytopenic Purpura in Children"
Acronym: ITP
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reham Elsayed Mohamed, Principal Investigator, Sohag University
Other Study IDs: SOH-Med--25-5-4MD
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: ITP - Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- investigate the potential association of single gene polymorphisms of CTLA-4 (SNPs; rs: 3087243) usi

SUMMARY:
the investigators aim in this study to investigate the potential association of single gene polymorphisms of CTLA-4 (SNPs; rs: 3087243) using real-time PCR in children with primary ITP.

DETAILED DESCRIPTION:
Primary immune thrombocytopenia (ITP) is an acquired autoimmune bleeding disorder characterized by isolated thrombocytopenia (platelet count < 100 × 109/L) in the absence of other etiologies. The incidence of the disease is approximately 2-10 per 100,000 adults each year, with a prevalence of 9-20 per 100,000 adults Auto antibody-mediated platelet destruction is the canonical mechanism of platelet destruction in ITP. Platelets coated by anti-glycoprotein (GP) autoantibodies are prematurely destroyed by macrophages via Fcγ receptors (FcγRs) in the reticuloendothelial system. Autoantibodies also accelerate platelet destruction through the induction of complement-dependent cytotoxicity (CDC) and platelet apoptosis Many studies have demonstrated that CD8+ cytotoxic T lymphocytes (CTLs) from peripheral blood or spleen of ITP patients can directly lyse platelets or induce platelet apoptosis through granzyme B and perforin. CTLs and anti-GP autoantibodies can induce the desialylation of platelet surface glycans, leading to premature platelet clearance.

The immune checkpoint pathways are critical modulators of the immune system, allowing immune response initiation and preventing autoimmunity onset. Immune checkpoints, including co-stimulation and co-inhibition signal pathways, are among the central mechanisms that regulate T-cell-mediated immune responses CTLA-4 production is strongly influenced by genetic factors. Single-nucleotide polymorphisms (SNPs) of the CTLA-4-encoding genes are involved in the pathogenesis of many autoimmune diseases such as systemic lupus erythematosus (SLE) and rheumatoid arthritis (RA) In recent years, it had been shown that thrombocytopenia was associated with the transcription level of CTLA4 and regulation of T-cell activation

ELIGIBILITY:
Inclusion criteria: approval to sign an informed written consent, patient with newly diagnosed ITP, patient age > 1 year and < 18 years and both sexes are included.

Exclusion criteria:

Refusal to sign an informed written consent, patient with persistent ITP, patient with chronic ITP, patient with secondary immune thrombocytopenia and patient age < 1 year or > 18 years

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. Full history taking.
  2. Through clinical examination.
  3. Laboratory investigations:
  a .Complete blood count with platelet indices: Mean Platelet Volume, Plateletcrit, platelet distribution width (MPV, PCT & PDW).
  b. Genotyping of rs3087243-related single-nucleotide polymorphism.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2027-06-04 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
investigate the potential association of single gene polymorphisms of CTLA-4 (SNPs; rs: 3087243) using real-time PCR in children with primary ITP. | Baseline